CLINICAL TRIAL: NCT04868838
Title: A Phase 2 Open-label Trial Evaluating the Efficacy and Safety of Daratumumab in Treatment of Patients With Active Lupus Nephritis
Brief Title: Daratumumab to Treat Active Lupus Nephritis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fernando Fervenza, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-010520
Record Dates: First submitted 2021-04-20; First posted 2021-05-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental): Subjects diagnosed with lupus nephritis will receive Daratumumab once weekly for 8 weeks and then once every 2 weeks for 8 additional does (+/- 4 days). Subjects will be followed for a total of 24 months (18 months after the last daratumumab administration).
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — 1800 mg administered by subcutaneous injection by manual push over approximately 3-5 minutes in the abdominal subcutaneous tissues in the left/right locations, alternating between individual doses.

SUMMARY:
The purpose of this research is to study the safety and efficacy of daratumumab in inducing complete or partial remission in patients with active lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Diagnosis of SLE according to current American College of Rheumatology (ACR) criteria.
* Renal biopsy confirming the diagnosis of active class III/IV (± class V) LN (based on International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003) within 12 months of enrollment.
* Proteinuria ≥ 500 mg over 24 hours.
* eGFR ≥ 30 ml/min/SA.
* Subjects should be able to give informed consent.

Exclusion Criteria:

* Pregnancy.
* Hepatitis B or C, HIV
* Anemia with Hgb < 8.0 g/dL.
* Thrombocytopenia with platelet count < 100'000.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication.
* Unable to provide consent.
* Patients receiving > 10 mg of oral prednisone or glucocorticoid equivalent if on corticosteroids for > 2 weeks (patients would be allowed to be on > 10 mg of prednisone or its oral equivalent as long as the duration is ≤ 2 weeks).
* Patients who had received immunosuppressive therapy including cyclosporine, tacrolimus or azathioprine in the last 3 months.
* Patients who have received cyclophosphamide in the last 6 months.
* Patients who received rituximab previously with CD20 count of zero at the time of enrollment.
* Patient are allowed to be on MMF at time of enrollment but no higher than total of 1500mg/day.
* For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 12 months after the last dose of study drug.
* For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study drug and agreement to refrain from donating sperm during this same period.
* Patients with diagnosis of glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of daratumumab in inducing complete(CR) or partial(PR) renal remission in patients with active class III or IV Lupus Nephritis | 12 months after first infusion of Daratumumab
  Complete Renal Response:- < 500 mg proteinuria/24 hours, Inactive urinary sediment (<10 RBC/HPF and absence of RBC casts), No greater than a 15% reduction in eGFR from enrollment
Efficacy of daratumumab in inducing complete(CR) or partial(PR) | 12 months after first infusion of Daratumumab
  Partial Renal Response: > 50% reduction in 24-hour proteinuria and proteinuria < 1g/24hr if baseline 24hr proteinuria, - ≤3 g/24hr and proteinuria ≤ 3 g/24hr if starting proteinuria > 3 g/24hrs. , Improved urinary sediment (>=50% reduction in RBC/HPF and absence of RBC casts), No greater than a 20% reduction in baseline eGFR

SECONDARY OUTCOMES:
Safety of daratumumab in patients with active class III/IV LN. | 24 months after first infusion of Daratumumab
  Incidence of major infections defined in the development of pneumonia, grade 3 urinary tract infection/pyelonephritis, sepsis, meningitis or anemia.
Improvement from proteinuria | Baseline, 6, 12, 18 and 24 months after first infusion of Daratumumab
  Change in proteinuria in milligrams (mg) per 24h
Change in hematuria. | Baseline,6, 12, 18 and 24 months after first infusion of Daratumumab
  Improvement in hematuria from baseline as measured by the urinalysis
Improvement in eGFR | Baseline, 6, 12, 18 and 24 months after first infusion of Daratumumab
  Improvement in eGFR measured using the chronic kidney disease epidemiology collaboration (CKD-EPI) Equation: eGFR (CKD-EPI) = 141 x min(Scr/k, 1)alpha x max(Scr/k,1)-1.209 x 0.993age x 1.018 (if patient is female) x 1.159 (if patient is black)
Change in ds-DNA | Baseline, 6, 12, 18 and 24 months after first infusion of Daratumumab
  Improvement in ds-DNA in International units per milliliter (IU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Plan pending

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials